CLINICAL TRIAL: NCT00284609
Title: "The Effect of Rehabilitation of Type 2 Diabetes Mellitus Versus Standard Outpatient Care." A Randomized Controlled Trial.
Brief Title: Rehabilitation of Type 2 Diabetes Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: National Board of Health, Denmark (Other Government); The Health and Care Committee, Copenhagen City Council (Unknown)
Responsible Party: Michael Røder, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: (KF) 01 287360; 2005-41-6000; MPU 39-2005
Record Dates: First submitted 2006-01-17; First posted 2006-02-01 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2009-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes,; rehabilitation,; quality of life,; glycaemic control,; lifestyle intervention,; patient education,; physical training,; group visits,; reminders
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Group based non-pharmacological rehabilitation
- 2 (Active Comparator)
  Interventions: Behavioral: Individual non-pharmacological rehabilitation

INTERVENTIONS:
Behavioral: Group based non-pharmacological rehabilitation — 6 x 1.5 hours education program in group classes taught by nurse, physiotherapist, dietitian and chiropodist.
  24 x 1.5 hours training program (both aerobic and anaerobic exercise) in group classes supervised by a physiotherapist.
  3 x 3 hours cooking sessions in group classes supervised by a dietitian.
  Intervention period: 6 month
  Arms: 1
Behavioral: Individual non-pharmacological rehabilitation — Individual counseling in Outpatient Clinic, including patient education, physical activity and diet instruction.
  4 x 1 hour with a diabetes nurse,
  3 x 0.5 hour with a dietitian and
  1 hour with a chiropodist.
  Intervention period: 6 month
  Arms: 2

SUMMARY:
The aim of this study is to investigate the effect of a new rehabilitation program of type 2 diabetes patients in a primary care center versus standard care in the outpatient Hospital Clinic.

DETAILED DESCRIPTION:
Type 2 diabetes is major and growing health care problem and is associated with premature mortality and increased morbidity. At the time of diagnosis half of the patients have cardiovascular, renal, ophthalmic or neurological disease. A recent Danish intervention study found a marked reduction in cardiovascular events and microvascular complications in a group of patients with type 2 diabetes and microalbuminuria using an intensive multifactorial pharmacologic intervention and lifestyle intervention (3). The achieved changes in lifestyle seems however to vanish after a short period. Lack of information, unawareness of the seriousness of the disease and lack of supervised training and insufficient follow-up may be of importance of the long-term outcome in these patients.

A total number of 180 patients with type 2 diabetes, will be randomized to the intervention group or to standard care.

This study tests an intensive intervention of lifestyle by a newly developed program of rehabilitation compared with routine standards in a randomized controlled design. Provided that a significant positive outcome is found, the non-pharmacologic treatment of type 2 diabetes could be optimized and inpatient hospitalization due to complications could be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 diabetes mellitus
* HgbA1c between 6,8 - 10,0%
* With or without one or more micro- and macrovascular or neurological complications.

Exclusion Criteria:

* HgbA1c < 6,8 and > 10,0 %
* Patients who have attended lifestyle intervention in the past year
* Patients who is planned to start treatment with insulin during intervention period
* Lack of motivation
* Patients with severe heart-, liver or kidney disease or incurable cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2006-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in HgbA1c (Glycemic control) | baseline, six month, one year, two years and three years

SECONDARY OUTCOMES:
fasting total cholesterol, triglycerides, HDL and LDL, | baseline, six month, one year, two years and three years
blood pressure, | baseline, six month, one year, two years and three years
weight, | baseline, six month, one year, two years and three years
waist circumference, | baseline, six month, one year, two years and three years
fitness test, | baseline, six month, one year, two years and three years
muscle strength test, | baseline, six month, one year, two years and three years
occurrence of complications, | baseline, six month, one year, two years and three years
inflammatory markers, | baseline, six month, one year, two years and three years
beta-cell function test (HOMA-test), | baseline, six month, one year, two years and three years
endothelia cell markers, | Not yet known
use of medication | baseline, six month, one year, two years and three years
cost-benefit. | Not yet known
Change in Quality of Life | baseline, six month, one year, two years and three years
Body mass index | baseline, six month, one year, two years and three years

CONTACTS AND LOCATIONS:
Overall Officials: Eva S Vadstrup, MD, Principal Investigator — Endocrine Section, Dept Internal Medicine I, Bispebjerg Hospital, University of Copenhagen; Michael Røder, DMSc, Study Director — Endocrine Section, Dept Internal Medicine I, Bispebjerg Hospital, University of Copenhagen
Locations (1):
- Endocrine Section, Dept Internal Medicine I, Bispebjerg Hospital, University of Copenhagen, Copenhagen, Copenhagen NV, Denmark

REFERENCES:
- [Background] Gaede P, Vedel P, Larsen N, Jensen GV, Parving HH, Pedersen O. Multifactorial intervention and cardiovascular disease in patients with type 2 diabetes. N Engl J Med. 2003 Jan 30;348(5):383-93. doi: 10.1056/NEJMoa021778. PMID 12556541
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Boule NG, Haddad E, Kenny GP, Wells GA, Sigal RJ. Effects of exercise on glycemic control and body mass in type 2 diabetes mellitus: a meta-analysis of controlled clinical trials. JAMA. 2001 Sep 12;286(10):1218-27. doi: 10.1001/jama.286.10.1218. PMID 11559268
- [Background] Boule NG, Kenny GP, Haddad E, Wells GA, Sigal RJ. Meta-analysis of the effect of structured exercise training on cardiorespiratory fitness in Type 2 diabetes mellitus. Diabetologia. 2003 Aug;46(8):1071-81. doi: 10.1007/s00125-003-1160-2. Epub 2003 Jul 10. PMID 12856082
- [Background] Krotkiewski M, Lonnroth P, Mandroukas K, Wroblewski Z, Rebuffe-Scrive M, Holm G, Smith U, Bjorntorp P. The effects of physical training on insulin secretion and effectiveness and on glucose metabolism in obesity and type 2 (non-insulin-dependent) diabetes mellitus. Diabetologia. 1985 Dec;28(12):881-90. doi: 10.1007/BF00703130. PMID 3912243
- [Background] Yeater RA, Ullrich IH, Maxwell LP, Goetsch VL. Coronary risk factors in type II diabetes: response to low-intensity aerobic exercise. W V Med J. 1990 Jul;86(7):287-90. PMID 2368376
- [Background] Wing RR. Physical activity in the treatment of the adulthood overweight and obesity: current evidence and research issues. Med Sci Sports Exerc. 1999 Nov;31(11 Suppl):S547-52. doi: 10.1097/00005768-199911001-00010. PMID 10593526
- [Background] Renders CM, Valk GD, Griffin SJ, Wagner EH, Eijk Van JT, Assendelft WJ. Interventions to improve the management of diabetes in primary care, outpatient, and community settings: a systematic review. Diabetes Care. 2001 Oct;24(10):1821-33. doi: 10.2337/diacare.24.10.1821. PMID 11574449
- [Background] Norris SL, Lau J, Smith SJ, Schmid CH, Engelgau MM. Self-management education for adults with type 2 diabetes: a meta-analysis of the effect on glycemic control. Diabetes Care. 2002 Jul;25(7):1159-71. doi: 10.2337/diacare.25.7.1159. PMID 12087014
- [Background] GESICA Investigators. Randomised trial of telephone intervention in chronic heart failure: DIAL trial. BMJ. 2005 Aug 20;331(7514):425. doi: 10.1136/bmj.38516.398067.E0. PMID 16061499
- [Background] Han TS, van Leer EM, Seidell JC, Lean ME. Waist circumference action levels in the identification of cardiovascular risk factors: prevalence study in a random sample. BMJ. 1995 Nov 25;311(7017):1401-5. doi: 10.1136/bmj.311.7017.1401. PMID 8520275
- [Background] Rexrode KM, Carey VJ, Hennekens CH, Walters EE, Colditz GA, Stampfer MJ, Willett WC, Manson JE. Abdominal adiposity and coronary heart disease in women. JAMA. 1998 Dec 2;280(21):1843-8. doi: 10.1001/jama.280.21.1843. PMID 9846779
- [Background] Lakka HM, Lakka TA, Tuomilehto J, Salonen JT. Abdominal obesity is associated with increased risk of acute coronary events in men. Eur Heart J. 2002 May;23(9):706-13. doi: 10.1053/euhj.2001.2889. PMID 11977996
- [Background] Bigaard J, Tjonneland A, Thomsen BL, Overvad K, Heitmann BL, Sorensen TI. Waist circumference, BMI, smoking, and mortality in middle-aged men and women. Obes Res. 2003 Jul;11(7):895-903. doi: 10.1038/oby.2003.123. PMID 12855760
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Derived] Vadstrup ES, Frolich A, Perrild H, Borg E, Roder M. Effect of a group-based rehabilitation programme on glycaemic control and cardiovascular risk factors in type 2 diabetes patients: the Copenhagen Type 2 Diabetes Rehabilitation Project. Patient Educ Couns. 2011 Aug;84(2):185-90. doi: 10.1016/j.pec.2010.06.031. Epub 2010 Aug 10. PMID 20702058
- [Derived] Vadstrup ES, Frolich A, Perrild H, Borg E, Roder M. Lifestyle intervention for type 2 diabetes patients: trial protocol of The Copenhagen Type 2 Diabetes Rehabilitation Project. BMC Public Health. 2009 May 29;9:166. doi: 10.1186/1471-2458-9-166. PMID 19480671